CLINICAL TRIAL: NCT04295005
Title: The Empagliflozin vs. DPP-4 Inhibitors and GLP-1 Receptor Agonists Cost of Care Study: a German Claims Data Analysis
Brief Title: A Study Based on Data From German Sick Funds That Looks at the Costs of Treatment of Type-2 Diabetic Patients With Empagliflozin vs. DPP-4 Inhibitors vs. GLP-1 Receptor Agonists
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0221
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- All patients who started an Empagliflozin therapy: All participants who met the inclusion criteria and none of the exclusion criteria of this study, who had at least two outpatient diagnoses and/or one inpatient diagnosis of Type 2 diabetes mellitus (T2DM) and received at least one outpatient prescription with Empagliflozin (EMPA) between 2015 - 2018 from the Gesellschaft für Qualität und Wirtschaftlichkeit bei Krankenkassen (GWQ) dataset.
  Interventions: Drug: Empagliflozin
- All patients who started a DPP-4 inhibitor (specifically Sitagliptin) therapy: All participants who met the inclusion criteria and none of the exclusion criteria of this study, who had at least two outpatient diagnoses and/or one inpatient diagnosis of Type 2 diabetes mellitus (T2DM) and received at least one outpatient prescription with Dipeptidyl peptidase 4 (DPP-4) inhibitor (DPP-4i) (specifically Sitagliptin) between 2015 - 2018 from the Gesellschaft für Qualität und Wirtschaftlichkeit bei Krankenkassen (GWQ) dataset.
  Interventions: Drug: DPP-4i
- All patients who started a GLP-1 receptor agonist therapy: All participants who met the inclusion criteria and none of the exclusion criteria of this study, who had at least two outpatient diagnoses and/or one inpatient diagnosis of Type 2 diabetes mellitus (T2DM) and received at least one outpatient prescription with Glucagon-like peptide-1 (GLP-1) receptor agonist (GLP-1-RA) between 2015 - 2018 from the Gesellschaft für Qualität und Wirtschaftlichkeit bei Krankenkassen (GWQ) dataset.
  Interventions: Drug: GLP-1-RA

INTERVENTIONS:
Drug: Empagliflozin — film coated tablet
  Groups: All patients who started an Empagliflozin therapy
Drug: DPP-4i — film coated tablets, specifically Sitagliptin
  Groups: All patients who started a DPP-4 inhibitor (specifically Sitagliptin) therapy
Drug: GLP-1-RA — subcutaneous injection or tablet
  Groups: All patients who started a GLP-1 receptor agonist therapy

SUMMARY:
Empagliflozin vs. Dipeptidyl Peptidase 4 (DPP-4) Inhibitors and Glucagon-like Peptide-1 Receptor Agonists (GLP-1-RA) Cost of Care Study: a German claims data analysis

ELIGIBILITY:
Inclusion Criteria:

* Continuous insurance by the sickness fund for the entire period (01/01/2014 - 31/12/2018; death of a patient is the only accepted exception from this rule)
* At least two outpatient T2DM diagnoses (ICD E11.-) in two different quarters and/or at least one inpatient T2DM diagnosis (ICD E11.-) in the period 01/01/2014 to 31/12/2016, but before or on index date (i.e. first Empagliflozin or DPP-4i /Sitagliptin prescription).
* At least one prescription of Empagliflozin or a DPP-4i /Sitagliptin in the inclusion period (01/01/2015 - 31/12/2016)

Exclusion Criteria:

* At least one prescription of a sodium glucose transporter 2 inhibitor (SGLT-2i), DPP-4i or GLP-1-RA in the baseline period (01/01/2014 - 31/12/2014)

  * During follow-up, patients will be censored if they switch to any SGLT-2i, DPP-4i or GLP-1-RA or initiate a concomitant use of any SGLT-2i, DPP-4i or GLP-1-RA (free or fixed-dose combinations).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes mellitus (T2DM) patients who have been treated with either Empagliflozin, DPP-4i /Sitagliptin or GLP-1-RA (new users only, at least one prescription).
Sampling Method: Probability Sample
Enrollment: 24500 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim, Ingelheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This retrospective study was to compare healthcare cost associated with different antidiabetic drug treatments among the incident users of Empagliflozin (EMPA), any Dipeptidyl peptidase 4 inhibitor (DPP-4i) (specifically Sitagliptin) or any Glucagon-like peptide-1 receptor agonist (GLP-1-RA), based on data covering 2015 - 2018 from Gesellschaft für Qualität und Wirtschaftlichkeit bei Krankenkassen (GWQ) dataset.
Pre-assignment Details: All subjects who strictly met all inclusion and none of the exclusion criteria were included in the study.
Period: Overall Study
Arm/Group | All Patients Who Started an Empagliflozin Therapy | All Patients Who Started a DPP-4 Inhibitor (Specifically Sitagliptin) Therapy | All Patients Who Started a GLP-1 Receptor Agonist Therapy
Started | 3285 | 19433 | 1747
Patients Who Started a Sitagliptin Therapy | 0 | 18382 | 0
Completed | 3285 | 19433 | 1747
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | All Patients Who Started an Empagliflozin Therapy | All Patients Who Started a DPP-4 Inhibitor (Specifically Sitagliptin) Therapy | All Patients Who Started a GLP-1 Receptor Agonist Therapy | Total
Number analyzed (Participants) | 3285 | 19433 | 1747 | 24465
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (11.0) | 63.3 (12.6) | 55.0 (12.0) | 62.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1110 | 7705 | 754 | 9569
  Male | 2175 | 11728 | 993 | 14896
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Direct Healthcare Cost
Description: The direct healthcare cost is reported, including inpatient cost, outpatient cost, medication cost, and total cost. Patients starting Empagliflozin (EMPA) versus either Dipeptidyl peptidase 4 inhibitor (DPP-4i), Sitagliptin (SITA) or Glucagon-like peptide-1 receptor agonist (GLP-1-RA) were matched 1:1 based on a propensity score using a nearest-neighbor matching algorithm without replacement and a maximum caliper of 0.001. The propensity scores were derived by logistic regression models estimating the probability of a patient belonging to the different treatment groups (three estimations: EMPA versus DPP-4i, EMPA versus SITA, and EMPA versus GLP-1-RA). The cost per observed patient year is calculated as the sum of the cost/ sum of the observed time [year] over all patients. Final values were rounded to the nearest digit.
Time Frame: Dataset included all adult persons, who were continuously insured between 01 january 2014 until 31 december 2018 (except for death), approximately a 4 year period.
Population: All eligible participants in this study, with non-missing outcome measures, and matched via propensity score adjusting for potential differences in patient characteristics and prior disease and treatment history among cohorts. The Dipeptidyl peptidase 4 inhibitor (DPP-4i) group and the Sitagliptin group are not mutually exclusive.
Measure: Mean (95% Confidence Interval); unit: Euro / patient-year
Groups:
- Empagliflozin (Matched to Dipeptidyl Peptidase 4 Inhibitor (DPP-4i)): Matched participants who met the inclusion criteria and none of the exclusion criteria of this study, who had at least two outpatient diagnoses and/or one inpatient diagnosis of Type 2 diabetes mellitus (T2DM) and received at least one outpatient prescription with Empagliflozin (EMPA) between 2015 - 2018 before this study start from the Gesellschaft für Qualität und Wirtschaftlichkeit bei Krankenkassen (GWQ) dataset.
  This cohort includes participants prescribed empagliflozin and who were matched to Dipeptidyl peptidase 4 inhibitor (DPP-4i) cohort via propensity score matching adjusting for potential differences in patient characteristics and prior disease and treatment history between the two cohorts.
- Dipeptidyl Peptidase 4 Inhibitor (DPP-4i) (Matched): Matched participants who met the inclusion criteria and none of the exclusion criteria of this study, who had at least two outpatient diagnoses and/or one inpatient diagnosis of Type 2 diabetes mellitus (T2DM) and received at least one outpatient prescription with Dipeptidyl peptidase 4 (DPP-4) inhibitor (DPP-4i) between 2015 - 2018 before this study start from the Gesellschaft für Qualität und Wirtschaftlichkeit bei Krankenkassen (GWQ) dataset.
  This cohort includes participants prescribed DPP-4i and who were matched to Empagliflozin cohort via propensity score matching adjusting for potential differences in patient characteristics and prior disease and treatment history between the two cohorts.
- Empagliflozin (Matched to Sitagliptin (SITA)): This cohort includes participants prescribed empagliflozin and who were matched to Sitagliptin (SITA) cohort via propensity score matching adjusting for potential differences in patient characteristics and prior disease and treatment history between the two cohorts.
- Sitagliptin (SITA) (Matched): Matched participants who met the inclusion criteria and none of the exclusion criteria of this study, who had at least two outpatient diagnoses and/or one inpatient diagnosis of Type 2 diabetes mellitus (T2DM) and received at least one outpatient prescription with Sitagliptin between 2015 - 2018 before this study start from the Gesellschaft für Qualität und Wirtschaftlichkeit bei Krankenkassen (GWQ) dataset.
  This cohort includes participants prescribed SITA and who were matched to Empagliflozin cohort via propensity score matching adjusting for potential differences in patient characteristics and prior disease and treatment history between the two cohorts.
- Empagliflozin (Matched to Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA)): This cohort includes participants prescribed empagliflozin and who were matched to Glucagon-like peptide-1 receptor agonist (GLP-1-RA) cohort via propensity score matching adjusting for potential differences in patient characteristics and prior disease and treatment history between the two cohorts.
- Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA) (Matched): Matched participants who met the inclusion criteria and none of the exclusion criteria of this study, who had at least two outpatient diagnoses and/or one inpatient diagnosis of Type 2 diabetes mellitus (T2DM) and received at least one outpatient prescription with Glucagon-like peptide-1 (GLP-1) receptor agonist (GLP-1-RA) between 2015 - 2018 before this study start from the Gesellschaft für Qualität und Wirtschaftlichkeit bei Krankenkassen (GWQ) dataset.
  This cohort includes participants prescribed GLP-1-RA and who were matched to Empagliflozin cohort via propensity score matching adjusting for potential differences in patient characteristics and prior disease and treatment history between the two cohorts.
Arm/Group | Empagliflozin (Matched to Dipeptidyl Peptidase 4 Inhibitor (DPP-4i)) | Dipeptidyl Peptidase 4 Inhibitor (DPP-4i) (Matched) | Empagliflozin (Matched to Sitagliptin (SITA)) | Sitagliptin (SITA) (Matched) | Empagliflozin (Matched to Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA)) | Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA) (Matched)
Number analyzed (Participants) | 3100 | 3100 | 3102 | 3102 | 1346 | 1346
Euro / patient-year
  Total | 4247 [3982 to 4566] | 7009 [6573 to 7445] | 4319 [4024 to 4614] | 6535 [6150 to 6920] | 4895 [4345 to 5445] | 6851 [6183 to 7518]
  Inpatient | 1455 [1230 to 1680] | 3040 [2698 to 3382] | 1486 [1260 to 1713] | 2806 [2491 to 3121] | 1546 [1099 to 1922] | 2094 [1552 to 2637]
  Outpatient | 853 [814 to 892] | 1280 [1197 to 1363] | 863 [824 to 902] | 1213 [1165 to 1260] | 917 [854 to 980] | 1181 [1103 to 1258]
  Medication | 1966 [1826 to 2107] | 2689 [2522 to 2855] | 1970 [1830 to 2110] | 2516 [2379 to 2653] | 2433 [2189 to 2677] | 3575 [3331 to 3819]
Statistical Analysis 1: Comparison: Empagliflozin (Matched to Dipeptidyl Peptidase 4 Inhibitor (DPP-4i)) vs Dipeptidyl Peptidase 4 Inhibitor (DPP-4i) (Matched); Total cost comparison; Test type: Other — Group differences in the costs incurred after treatment initiation were evaluated based on an incremental cost approach using the Bang and Tsiatis estimator with possibly censored data; p < 0.001, Bang and Tsiatis
Statistical Analysis 2: Comparison: Empagliflozin (Matched to Sitagliptin (SITA)) vs Sitagliptin (SITA) (Matched); Total cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis
Statistical Analysis 3: Comparison: Empagliflozin (Matched to Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA)) vs Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA) (Matched); Total cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis
Statistical Analysis 4: Comparison: Empagliflozin (Matched to Dipeptidyl Peptidase 4 Inhibitor (DPP-4i)) vs Dipeptidyl Peptidase 4 Inhibitor (DPP-4i) (Matched); Inpatient cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis
Statistical Analysis 5: Comparison: Empagliflozin (Matched to Sitagliptin (SITA)) vs Sitagliptin (SITA) (Matched); Inpatient cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis
Statistical Analysis 6: Comparison: Empagliflozin (Matched to Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA)) vs Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA) (Matched); Inpatient cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.126, Bang and Tsiatis
Statistical Analysis 7: Comparison: Empagliflozin (Matched to Dipeptidyl Peptidase 4 Inhibitor (DPP-4i)) vs Dipeptidyl Peptidase 4 Inhibitor (DPP-4i) (Matched); Outpatient cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis
Statistical Analysis 8: Comparison: Empagliflozin (Matched to Sitagliptin (SITA)) vs Sitagliptin (SITA) (Matched); Outpatient cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis
Statistical Analysis 9: Comparison: Empagliflozin (Matched to Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA)) vs Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA) (Matched); Outpatient cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis
Statistical Analysis 10: Comparison: Empagliflozin (Matched to Dipeptidyl Peptidase 4 Inhibitor (DPP-4i)) vs Dipeptidyl Peptidase 4 Inhibitor (DPP-4i) (Matched); Medication cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis
Statistical Analysis 11: Comparison: Empagliflozin (Matched to Sitagliptin (SITA)) vs Sitagliptin (SITA) (Matched); Medication cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis
Statistical Analysis 12: Comparison: Empagliflozin (Matched to Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA)) vs Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA) (Matched); Medication cost comparison; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, Bang and Tsiatis

2. Primary Outcome: Healthcare Resource Utilization
Description: Healthcare resource utilization includes hospitalizations, hospital stays. outpatient visits, and rehabilitation stays.
Time Frame: as for outcome 1
Population: Relevant data for the outcome measure were not collected in the GMQ dataset because GWQ´s quality assurance decided not to integrate several sub-datasets into GWQ´s dataset due to heterogeneity and low coding-quality of out-patient diagnoses and high variability in size, structure, and quality of specific items in individual sickness funds data.
Arm/Group | Empagliflozin (Matched to Dipeptidyl Peptidase 4 Inhibitor (DPP-4i)) | Dipeptidyl Peptidase 4 Inhibitor (DPP-4i) (Matched) | Empagliflozin (Matched to Sitagliptin (SITA)) | Sitagliptin (SITA) (Matched) | Empagliflozin (Matched to Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA)) | Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA) (Matched)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Indirect Healthcare Costs (Including Indirect Costs of Days Absent From Work)
Description: Indirect healthcare costs (including indirect costs of days absent from work) includes indirect costs for hospitalization, outpatient visits, absent from work, and rehabilitation stays.
Time Frame: as for outcome 1
Population: as for outcome 2
Arm/Group | Empagliflozin (Matched to Dipeptidyl Peptidase 4 Inhibitor (DPP-4i)) | Dipeptidyl Peptidase 4 Inhibitor (DPP-4i) (Matched) | Empagliflozin (Matched to Sitagliptin (SITA)) | Sitagliptin (SITA) (Matched) | Empagliflozin (Matched to Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA)) | Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA) (Matched)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: This is a non-interventional study using electronic health care records, with data retrieved from Gesellschaft für Qualität und Wirtschaftlichkeit bei Krankenkassen (GWQ). The adverse events were not planned to be collected and reported. The "0" in the All-Cause Mortality, Serious Adverse Events, and Other (non-serious) Adverse Events sections refers to "not applicable".
Arm/Group | All Patients Who Started an Empagliflozin Therapy | All Patients Who Started a DPP-4 Inhibitor (Specifically Sitagliptin) Therapy | All Patients Who Started a GLP-1 Receptor Agonist Therapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Relevant data for the outcome measure were not collected in the GMQ dataset. The general reason for missing data in GWQ´s dataset is insufficient data quality. First, coding-quality of out-patient diagnoses in Germany is heterogenous and generally low. Second, data from GWQ´s individual sickness funds highly differ in size, structure, and quality of specific items. Due to this, GWQ´s quality assurance decided not to integrate several sub-datasets into GWQ´s dataset.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT04295005/Prot_SAP_000.pdf